CLINICAL TRIAL: NCT03135184
Title: HDL Acute Lipid Optimization in Homozygous Familial Hypercholesterolemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: HDL Therapeutics (Industry)
Collaborators: MedStar Heart and Vascular Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HALO-FH
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Homozygous Familial Hypercholesterolemia; HoFH
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Prospective, unblinded, interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- HDL Therapeutics PDS-2™ System (Experimental): Serial infusions of autologous selectively delipidated HDL/preβ enriched plasma following use of HDL Therapeutics PDS-2™ System
  Interventions: Device: HDL Therapeutics PDS-2 System

INTERVENTIONS:
Device: HDL Therapeutics PDS-2 System — Delipidation of plasma HDL to reduce coronary atheroma

SUMMARY:
Assess the effect on coronary atheroma of serial infusions of autologous selectively delipidated HDL/preβ enriched plasma following use of HDL Therapeutics PDS-2™ System

DETAILED DESCRIPTION:
The PDS-2™ System is intended to reduce coronary atheroma in patients with Homozygous Familial Hypercholesterolemia (HoFH). Subjects will receive serial infusions of autologous selectively delipidated HDL/preβ enriched plasma following use of HDL Therapeutics' PDS-2 System.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of Homozygous Familial Hypercholesterolemia (HoFH) due to a defect in the LDL receptor, or the identification of a defect in apoB-100, or a gain of function of PCSK9, or a genetic defect resulting in the HoFH clinical phenotype
* No other condition that would preclude the subject from successfully completing the series of plasmapheresis visits in the investigator's opinion
* At least one (1) coronary artery study segment will be identified for each subject and all will remain constant throughout the study. The qualifying study segment(s) will have 20% to 40% stenosis.

Key Exclusion Criteria:

* Planned change in current lipid lowering therapy
* Use of oral anticoagulants, unless the dose has been stable for 4 weeks
* LDL or plasma apheresis within 1 week prior to enrollment and through 8-week primary endpoint
* New York Heart Association (NYHA) class III or IV or last known left ventricular ejection fraction < 30%
* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 3 months of enrollment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Change in coronary atheroma | 2 months
  Assessed by coronary imaging in study coronary artery segments following serial infusions of autologous selectively delipidated HDL/preβ enriched plasma following use of HDL Therapeutics PDS-2™ System as compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center (CSMC), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No